CLINICAL TRIAL: NCT03902925
Title: Pain During Pars Plana Vitrectomy Comparing Peribulbar Anesthesia Versus Sub-tenon Injection Plus Topical Jelly Anesthesia
Brief Title: Pain During Pars Plana Vitrectomy With Sub-tenon Anesthesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jefferson Augusto Santana Ribeiro, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST anesthesia for PPV
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Retinal Disease; Diabetic Retinopathy; Maculopathy
Keywords: vitrectomy; anesthesia; retinal disease; Pain; diabetic retinopathy; maculopathy
MeSH Terms: conditions — Retinal Diseases; Diabetic Retinopathy; Macular Degeneration; Pain | interventions — Lidocaine; Gels; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Sub-tenon plus lidocaine jelly (Experimental): Patients are going to be submitted to lidocaine 2% jelly topical anesthesia for 5 minutes then to sub-tenon injection of 2-4 ml of ropivacaine 10% previous to 23 G pars plana vitrectomy.
  Interventions: Procedure: Topical lidocaine 2% jelly plus sub-tenon ropivacaine 10% injection
- Group 2- peribulbar (Active Comparator): Patients are going to be submitted to peribulbar injection of 4-6 ml of ropivacaine 10% previous to 23 G pars plana vitrectomy.
  Interventions: Procedure: Peribulbar injection

INTERVENTIONS:
Procedure: Topical lidocaine 2% jelly plus sub-tenon ropivacaine 10% injection — Lidocaine 2% jelly applied to conjunctival fornices for 5 minutes then injection of 2-4 ml of ropivacaine 10% in the sub-tenon space with a blunt cannula through a temporal inferior incision
  Arms: Group 1- Sub-tenon plus lidocaine jelly
Procedure: Peribulbar injection — Peribulbar injection of 4-6 ml of ropivacaine 10%
  Arms: Group 2- peribulbar

SUMMARY:
Vitreoretinal surgery has evolved to less invasive procedures, and it is used to treat a wide range of diseases. So anesthesia for vitreoretinal procedures has evolved, promoting adequate analgesia while reducing risks to the patient. In the present study two types of procedures for anesthesia during vitreoretinal surgery are evaluated regarding the pain referred by the patient during the whole procedure: peribulbar anesthesia versus sub-tenon injection plus topical jelly anesthesia. Through the comparative analysis of the pain scale of the two groups it is expected that the two modalities present the same anesthetic efficacy, showing that the methods used may be equivalent.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have the diagnosis of epiretinal membrane, macular hole, complication of diabetic retinopathy such as vitreous hemorrhage or traction retinal detachment or other vitreomacular diseases that require treatment by pars plana vitrectomy.

Exclusion Criteria:

* Previous pars plana vitrectomy in the studied eye.
* Previous scleral buckle surgery
* Uncontrolled arterial hypertension
* Any ocular surgery performed in the studied eye in the previous three months
* Medical or psychological condition that preclude study adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Pain score | Once 30 minutes after the end of the vitrectomy surgery
  Pain score referred by the patient measured with a Visual Analogue Scale (VAS). The VAS consists of ruler with 100 cm in length and scale from 0 to 100, where the numbers of this one are visible only in the side of the examiner. It is constructed from a metal ruler with a total length of one meter, supported by two transparent acrylic side supports and a sliding and movable metal weight on the metallic part of the ruler.
  Before the measurement of pain, the examiner will explain to the patients the functioning of the VAS. Each patient will be encouraged to pass the marker along the scale, with the help of the examiner. It will be made clear to him that point "0" is the point of the scale which represented "no pain", what is considered the better outcome, and point "100" corresponded to the most intense pain he could feel. The patient will be asked about: Intraoperative pain - the intensity of pain throughout the procedure.

SECONDARY OUTCOMES:
Surgical complications | Once At the end of vitrectomy surgery
  Surgical complications referred by the surgeon during vitrectomy

OTHER OUTCOMES:
Duration of surgery | Once At the end of vitrectomy surgery
  Duration of vitrectomy in minutes
Anesthetic medications | Once during the vitrectomy surgery
  Other anesthetic medication for controlling pain administered during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson AS Ribeiro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Medicine - Clinical Hospital, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We intend to have patient data stored but not individually available for researches at other sites in order to preserve anonymity of the patient.

REFERENCES:
- [Background] Tang S, Lai P, Lai M, Zou Y, Li J, Li S. Topical anesthesia in transconjunctival sutureless 25-gauge vitrectomy for macular-based disorders. Ophthalmologica. 2007;221(1):65-8. doi: 10.1159/000096526. PMID 17183205
- [Background] Stevens JD, Foss AJ, Hamilton AM. No-needle one-quadrant sub-tenon anaesthesia for panretinal photocoagulation. Eye (Lond). 1993;7 ( Pt 6):768-71. doi: 10.1038/eye.1993.180. PMID 8119430
- [Background] Spaeth G. Ophthalmic Surgery, Principles and Practice. Third Edition. Saunders, Philadelphia, 2003.
- [Background] Sousa FAEF, Silva JA. Avaliação e mensuração da dor em contextos clínicos e de pesquisa. Rev. Dor, 2004;5(4):408-429.
- [Background] Roman SJ, Chong Sit DA, Boureau CM, Auclin FX, Ullern MM. Sub-Tenon's anaesthesia: an efficient and safe technique. Br J Ophthalmol. 1997 Aug;81(8):673-6. doi: 10.1136/bjo.81.8.673. PMID 9349156
- [Background] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Background] Rao GP, Wong D, Groenewald C, McGalliard JN, Jones A, Ridges PJ. Local anaesthesia for vitreoretinal surgery: a case-control study of 200 cases. Eye (Lond). 1998;12 ( Pt 3a):407-11. doi: 10.1038/eye.1998.96. PMID 9775241
- [Result] Theocharis IP, Alexandridou A, Tomic Z. A two-year prospective study comparing lidocaine 2% jelly versus peribulbar anaesthesia for 25G and 23G sutureless vitrectomy. Graefes Arch Clin Exp Ophthalmol. 2007 Sep;245(9):1253-8. doi: 10.1007/s00417-007-0556-y. Epub 2007 Mar 7. PMID 17342504